CLINICAL TRIAL: NCT00591994
Title: Tinnitus Treatment With Piribedil Guided by Acoustic Otoemissions and Electrocochleography
Acronym: piribedil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Medicina de Valenca (Other)
Responsible Party: Andréia Aparecida de Azevedo, M.D., OTOSUL
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: OTOSUL 01/2007; FMV 01/2006
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2007-12

CONDITIONS: Tinnitus
Keywords: tinnitus; piribedil; acoustic otoemissions; ECoG
MeSH Terms: conditions — Tinnitus | interventions — Piribedil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: piribedil — 50 mg once a day, after lunch 3 month therapy

SUMMARY:
Tinnitus is defined as the perception of sound in the absence of a external source. About 15 % of the population is believed to experience tinnitus and for about 20 % of them it may become a very serious problem. Total comprehension of tinnitus pathophysiology has not yet been achieved, but modern theories focus in brain hyperactivity following inner ear damage, with involvement of various neurotransmitters. Piribedil,a dopamin agonist, has been used to treat tinnitus, focusing in dopamine release, which is inhibitory. Electrophysiological methods,like acoustic otoemissions and electrocochleography may reveal the changes in peripherical and central auditory pathways and help to choose the specific patients who could benefit from piribedil treatment.

ELIGIBILITY:
Inclusion Criteria:

* tinnitus for more than 6 months
* THI > 38
* no central acting drugs in the last 6 months
* tympanogram type A-n

Exclusion Criteria:

* vascular and muscular tinnitus
* concomitant TMJ disorders
* abnormal otoscopy
* mixed and conductive hearing losses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-11; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
THI - Tinnitus Handicap Inventory | Months 3 and 6

SECONDARY OUTCOMES:
VAS - Visual Analog Scale | Months 3 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo R Figueiredo, M.D.,M.Sc, Study Chair — Faculdade de Medicina de Valença; Andréia A Azevedo, M.D., Principal Investigator — Otosul -Otorrinolaringologia Sul-Fluminense
Locations (1):
- OTOSUL,Otorrinolaringologia Sul-Fluminense, Volta Redonda, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] de Azevedo AA, Langguth B, de Oliveira PM, Rodrigues Figueiredo R. Tinnitus treatment with piribedil guided by electrocochleography and acoustic otoemissions. Otol Neurotol. 2009 Aug;30(5):676-80. doi: 10.1097/MAO.0b013e3181ab8fd5. PMID 19574947